CLINICAL TRIAL: NCT03183232
Title: γδ T Cell Immunotherapy for Treatment of Lung Cancer
Brief Title: Safety and Efficiency of γδ T Cell Against Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: Jinan University Guangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Gd T cell and lung Ca
Record Dates: First submitted 2017-06-08; First posted 2017-06-12 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Lung Cancer
Keywords: Immunotherapy, γδ T Cell, Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Cryosurgery; Electroporation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): In this group, the patients will receive under CT Cryosurgery or IRE surgery to control the local tumor
  Interventions: Procedure: Cryosurgery or IRE surgery
- Group B (Experimental): In this group, the patients will receive multiple high-activity γδ T cell immunotherapies. The check indexes are CT scan and blood tests (including tumor markers, lymphocyte subsets and circulating tumor cell)
  Interventions: Biological: γδ T cell
- Group C (Experimental): In this group, the patients will receive multiple high-activity γδ T cell immunotherapies and Cryosurgery or IRE surgery
  Interventions: Other: γδ T cells/ A Cryosurgery or IRE

INTERVENTIONS:
Procedure: Cryosurgery or IRE surgery — Cryosurgery or IRE surgery will be used in local tumor
  Arms: Group A
Biological: γδ T cell — γδ T cells will be used against Lung Cancer
  Arms: Group B
Other: γδ T cells/ A Cryosurgery or IRE — Combination γδ T cell and Cryosurgery or IRE surgery will be used in Lung Cancer
  Arms: Group C

SUMMARY:
In this study, effects of γδT cells on human Lung Cancer in combination with tumor reducing surgery, for example, cryosurgery going to be investigated

DETAILED DESCRIPTION:
Lung tumor will be removed using tumor reducing surgery such as cryosurgery. PBMC of the patient will be separated from peripheral blood. After making them potential cancer killer γδ T Cell and DC-CIK, they will be infused to the patients as an immunotherapy treatment.

NOTE: Originally, our designed proposal was to use autologous PBMCs from cancer patients to ex vivo expand Vγ9Vδ2-T cells, and then perform adoptive transfer therapy. However, PBMCs of majority of cancer patients could not be effectively expanded, including cell number, cell purity and cell function could not meet the requirements of reinfusion. Meanwhile, those patients could not tolerate 100ml of blood drawing for culture every 2 ~ 3 weeks.

Therefore, we submitted new clinical study application to the ethical committee of the Fuda Hospital affiliated with Jinan University (Guangzhou, PR. China) by changing the autologous protocol with the allogeneic protocol. After the allogeneic protocol was approved, we adapted allogeneic cells instead of autologous in our subsequentially clinical study.

ELIGIBILITY:
Inclusion Criteria:

Age: 18-75 Karnofsky performance status >50 Diagnosis with Lung Cancer based on histology or the current accepted radiological measures Classification tumor,nodes,metastasis-classification(TNM) stage: Ⅱ,Ⅲ,Ⅳ Will receive cryosurgery, IRE, gd T cells Life expectancy: Greater than 3 months Ability to understand the study protocol and a willingness to sign a written informed consent document

Exclusion Criteria:

Patients with other kinds of cancer History of coagulation disorders or anemia Patients with heart disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Relief degree of tumors | 3 months
  It will be evaluated by the Response Evaluation Criteria in Solid Tumors
Progress free survival（PFS) | 1 year
Overall survival（OS） | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jibing Chen, PhD, Principal Investigator — Biological treatment center in Fuda cancer hospital Guangzhou, Guangdong, China, 510000
Locations (1):
- Biotherapy center in Fuda cancer hospital, Guangzhou, Guangdong, China